CLINICAL TRIAL: NCT04798157
Title: Role of Transcranial Doppler (TCD) in Children With Hemoglobinopathies
Brief Title: Transcranial Doppler in Children With Hemoglobinopathies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Elbadry Mohamed, teaching assistant , faculty of medicine , Sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-03-04
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Hemoglobinopathies
MeSH Terms: conditions — Hemoglobinopathies | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Hemoglobinopathies (Experimental): children from 2-18 years old , diagnosed to have hemoglobinopathy disease
  Interventions: Radiation: transcranial doppler

INTERVENTIONS:
Radiation: transcranial doppler — Transcranial Doppler ultrasonography will be done using the ultrasound machine by placing a transducer over the relatively thinner temporal and occipital bones in order to visualize and evaluate the velocities at the circle of Willis.

SUMMARY:
Transcranial Doppler ultrasonography (TCD) is a noninvasive, portable technique for evaluating the intracranial vasculature.

TCD ultrasonography is performed placing a low frequency (≤ 2 MHz) transducer on the scalp of the patient, in order to visualize the intracranial arterial vessels through specific acoustic windows, where bone is thinner, and evaluate cerebral blood flow velocity (CBFV) .

Patients diagnosed to have hemoglobinopathy conditions with its most common forms thalassemia and sickle cell disease manifest both biochemical and clinical evidence of hypercoagulability conditions include deep venous thrombosis, pulmonary emboli and recurrent arterial occlusion .

Cerebrovascular accidents can be identified using transcranial Doppler ultrasonography which enables evaluation of cerebral artery blood flow velocity with a sensitivity of 90% and specificity of 100 % when compared with cerebral angiography .

According to the stroke prevention trial in sickle cell anemia (STOP) study ,TCDs were classified based on blood velocity in the circle of Willis, expressed as time averaged mean of the maximum velocity (TAMMV). Children with abnormal, high velocities (>200cm/s) were at increased risk of stroke, which was reduced by 90% after starting regular blood transfusions. TAMMVs less than 170cm/s were classified as normal with annual TCD scanning recommended, whereas velocities between 170 and 200cm/s were called conditional, and followed up more closely without starting transfusion.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with hemoglobinopathies

Exclusion Criteria:

* Children before two years old .
* Hemoglobinopathy patients more than 18 years .
* Uncooperative patients .

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Changes in the blood flow velocities at the circle of Willis | At procedure exam time
  The children will be be subjected to Transcranial Doppler (TCD ) , and velocity indices will be obtained , the subjects will be classified according the TAMMV (time average mean maximum velocities ) into high risk group with TAMMV > 200 cm/sec , and normal group <170 cm/sec , and conditional group with TAMMV 170-200 cm/sec .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E. Mohamed, ass. teacher, Principal Investigator — Faculty of medicine Sohag university

IPD SHARING:
Plan to Share IPD: No